CLINICAL TRIAL: NCT01604785
Title: Low-dose Propofol for Abortive Therapy of Pediatric Migraine in the Emergency Department
Brief Title: Low-dose Propofol for Pediatric Migraine
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Garth Meckler, Associate Professor, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Meckler01
Record Dates: First submitted 2012-05-22; First posted 2012-05-24 (Estimated); Results first posted 2018-12-31 (Actual); Last update posted 2018-12-31 (Actual); Status verified 2018-12

CONDITIONS: Migraine Headache
Keywords: Migraine Headache; Pediatric
MeSH Terms: conditions — Migraine Disorders | interventions — Propofol; Anti-Inflammatory Agents, Non-Steroidal; Dopamine Antagonists

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental Treatment Group (Experimental): Propofol at subanesthetic dose via IV push
  Interventions: Drug: Propofol
- Standard Treatment Group (Active Comparator): Metaclopramide in combination with ketorolac and diphenhydramine via IV infusion
  Interventions: Drug: Standard Treatment

INTERVENTIONS:
Drug: Propofol — Sub-anesthetic dose propofol: 0.25 mg/kg IV push to maximum dose of 30mg q5 minutes to a maximum of 5 doses
  Other Names: Diprivan
  Arms: Experimental Treatment Group
Drug: Standard Treatment — Ketorolac, Diphenhydramine and Metoclopramide
  Other Names: NSAIDs / Dopamine Antagonists
  Arms: Standard Treatment Group

SUMMARY:
Propofol, a general anesthetic, has been suggested to be effective for the treatment of migraine headaches in adults when used in subanesthetic doses (lower doses than those used for anesthesia or sedation). Initial retrospective review of the investigators experience with propofol for migraine in children suggests that it is safe and may be more effective than standard treatments used in the emergency department. The investigators retrospective series had a small subject population and a larger study is needed to compare propofol to current available treatments.

Standard treatment currently consists of a "cocktail" of medications that include anti-nausea medicines (metoclopramide and diphenhydramine) and an analgesic (ketorolac) as well as intravenous fluids. Subjects assigned to the experimental group (Propofol) will receive the same intravenous fluids and up to five doses of propofol. All subjects will undergo assessment of their pain (self-rated on a scale from 0-10) before and after treatment. Post-visit clinical data will be collected from the subject's medical record and subjects will be called by telephone 24-48 hours after discharge from the emergency department to ask how they are doing and whether they required any additional treatments such as home medications or by other medical professionals other than OHSU.

DETAILED DESCRIPTION:
There has been little advancement in abortive migraine therapies in recent decades, and few proven treatments exist for acute migraine, particularly in children. Propofol, a general anesthetic, has been suggested to be effective for the treatment of migraine headaches in adults when used in subanesthetic doses (lower doses than those used for anesthesia or sedation). Initial retrospective review of the investigators experience with propofol for migraine in children suggests that it is safe and may be more effective than standard treatments used in the emergency department. The investigators retrospective series had a small subject population and a larger study is needed to compare propofol to current available treatments.

All subjects presenting to the pediatric emergency department with signs/symptoms of migraine headache will be screened for the study. Subjects who are eligible will be provided information about the study and consent/assent forms from a member of the research team, and asked whether they are interested in participating.

All study subjects will receive acetaminophen (Tylenol) or ibuprofen (Motrin) for their headache if they have not already tried these first-line treatments at home; those with persistent symptoms requiring further treatment who consent to participate in the study will be randomized to receive either standard treatment or propofol. Standard treatment currently consists of a "cocktail" of medications that include anti-nausea medicines (metoclopramide and diphenhydramine) and an analgesic (ketorolac) as well as intravenous fluids. Subjects assigned to the experimental group (Propofol) will receive the same intravenous fluids and up to five doses of propofol. All subjects will undergo assessment of their pain (self-rated on a scale from 0-10) before and after treatment. During treatment they will have close monitoring of their vital signs. No additional laboratory tests or procedures are involved. Post-visit clinical data will be collected from the subject's medical record and subjects will be called by telephone 24-48 hours after discharge from the emergency department to ask how they are doing and whether they required any additional treatments such as home medications or by other medical professionals other than OHSU.

The study data will be presented in summary tables that outline subjects' clinical presentation prior to treatments, and response to study drug during their visit. The main variables of interest include effectiveness (determined as a reduction in self-reported pain score), length of stay in the pediatric emergency department, recurrent headache requiring emergency treatment within 24 hours and whether any adverse effects occur. These will be compared between the 2 study groups with basic statistics.

ELIGIBILITY:
Inclusion Criteria:

* Children 7-18 years of age
* Acute Migraine Headache

Exclusion Criteria:

* Head Trauma
* CNS infection
* CNS tumor
* Previous CNS surgery or device

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 74 (Actual)
Dates: Start 2012-11; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Garth D Meckler, MD, MSHS, Principal Investigator — Oregon Health and Science University; David Sheridan, MD, Study Director — sheridda@ohsu.edu
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental Treatment Group: Propofol at subanesthetic dose via IV push
  Propofol: Sub-anesthetic dose propofol: 0.25 mg/kg IV push to maximum dose of 30mg q5 minutes to a maximum of 5 doses
  Total enrollment = 37 subjects
- Standard Treatment Group: Metaclopramide in combination with ketorolac and diphenhydramine via IV infusion
  Standard Treatment: Ketorolac, Diphenhydramine and Metoclopramide
  Total enrollment = 37 subjects
Period: Overall Study
Arm/Group | Experimental Treatment Group | Standard Treatment Group
Started | 37 | 37
Completed | 30 | 36
Not Completed | 7 | 1
Not completed — Repeat Visits Not Included in Analysis | 7 | 1

BASELINE CHARACTERISTICS:
Population: 1 patient excluded for repeat visit from ST arm 7 patients excluded for repeat visit from Experimental arm
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental Treatment Group | Standard Treatment Group | Total
Number analyzed (Participants) | 30 | 36 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.6 (2.1) | 14.6 (3.0) | 14.6 (2.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 28 | 49
  Male | 9 | 8 | 17
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30 | 36 | 66

OUTCOME MEASURES:

1. Primary Outcome: Change in Self-Assessed Pain
Description: Percent pain change after initial treatment using 10 point VAS scale
Time Frame: 15 minutes after administration
Measure: Number; unit: percentage change
Groups:
- Experimental Treatment Group: Propofol at subanesthetic dose via IV push
  Propofol: Sub-anesthetic dose propofol: 0.25 mg/kg IV push to maximum dose of 30mg q5 minutes to a maximum of 5 doses
  Total enrollment = 30 subjects
- Standard Treatment Group: Metaclopramide in combination with ketorolac and diphenhydramine via IV infusion
  Standard Treatment: Ketorolac, Diphenhydramine and Metoclopramide
  Total enrollment = 36 subjects
Arm/Group | Experimental Treatment Group | Standard Treatment Group
Number analyzed (Participants) | 30 | 36
percentage change | 51 | 59

2. Secondary Outcome: Rebound Headache at 24 Hour Follow-up Phone Call
Description: Percentage of subjects reporting recurrence of headache with pain greater than at time of discharge from Emergency Department
Time Frame: 24 hours
Population: Percentage of participants
Measure: Number; unit: Percentage of subjects reporting rebound
Arm/Group | Experimental Treatment Group | Standard Treatment Group
Number analyzed (Participants) | 30 | 36
Percentage of subjects reporting rebound | 25 | 66.7

3. Secondary Outcome: Emergency Department Length of Stay
Description: Length of stay from administration of medication to Emergency Department discharge in minutes
Time Frame: Duration of stay in Emergency Department in Minutes
Measure: Median (Full Range); unit: Minutes
Arm/Group | Experimental Treatment Group | Standard Treatment Group
Number analyzed (Participants) | 30 | 36
Minutes | 79 [22 to 460] | 111 [42 to 630]

ADVERSE EVENTS:
Arm/Group | Experimental Treatment Group | Standard Treatment Group
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/36
Other Adverse Events (participants affected / at risk) | 1/30 | 3/36
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental Treatment Group (N=30) | Standard Treatment Group (N=36)
Extrapyramidal Symptoms (Nervous system disorders) | 0 (0) | 3 (3) — Extrapyramidal symptoms
Hypoxemia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Transient self-resolved hypoxia to 89%

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No